CLINICAL TRIAL: NCT04392999
Title: A Pilot Study Comparing Intra-articular Corticosteroid Injections to Platelet Rich Plasma (PRP) as a Treatment for Cervical Facetogenic Pain
Brief Title: Intra-articular Corticosteroid Injections to Platelet Rich Plasma (PRP) for Cervical Facetogenic Pain
Acronym: PRICE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ELPRP01
Record Dates: First submitted 2020-04-30; First posted 2020-05-19 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Cervical Pain
Keywords: cervical pain; neck pain; platelet rich plasma; PRP
MeSH Terms: conditions — Neck Pain | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Eligible participants who consent to study participation will be randomized to one of two groups: PRP injections, or corticosteroid injections.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants as well as the individuals collecting and analyzing outcome data will be blinded. The Primary Investigator, who is also the physician delivering the study compound, will not be blinded but will have no role in data collection or analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma (Experimental): One time injection of 1.5-6cc of platelet rich plasma prepared from a blood sample into cervical facet joints. There is no trade/generic name
  Interventions: Drug: Intraarticular platelet rich plasma cervical facet injection
- Dexamethasone Sodium Phosphate (Active Comparator): Corticosteroid: 0.5 cc saline and 0.5cc of 10 mg/mL dexamethasone per facet joint (up to 6 mL total volume for 4 facet injections)
  Interventions: Drug: Corticosteroid injection

INTERVENTIONS:
Drug: Intraarticular platelet rich plasma cervical facet injection — Injection of PRP into the cervical facet joints.
  Other Names: PRP injection
  Arms: Platelet Rich Plasma
Drug: Corticosteroid injection — Injection of corticosteroid into the cervical facet joints.
  Arms: Dexamethasone Sodium Phosphate

SUMMARY:
Chronic neck pain, either after trauma (e.g. whiplash injury) or due to arthritis, is a significant issue for many Canadians. Steroid injections into the small joints of the neck can provide temporary pain relief, but patients require repeat injections every few months. The investigator will assess whether a different type of injection (platelet-rich plasma, PRP) can provide enhanced and longer-lasting pain relief compared to steroid. PRP is made from the patient's own blood but contains higher levels of components that promote healing. Patients with neck pain will receive either an injection of steroid or PRP into the small joints of the neck, but they won't know which one they are getting. After the injection they will be contacted to answer questions about their pain and function, up to 12 months after injection. The goal of this study is to determine if PRP is a viable alternative to current treatments to help reduce chronic neck pain and improve function after a whiplash injury. PRP may be a more permanent treatment for chronic neck pain which could reduce the need for repeated injections, thus reducing health care costs and wait times.

DETAILED DESCRIPTION:
The project utilizes a randomized control trial design. Ethics approval was obtained from the Western Research Ethics Board. Participants with chronic neck pain will be recruited from the SJHC Pain Clinic.

Eligible candidates who consent to study participation will be block randomized using randomizer.org into two groups (A or B). All patients will be blinded both before and after injections as to which therapy they receive. Group A will receive an intra-articular (IA) injection of autologous PRP (0.5 mL per level) and Group B will receive IA injections of corticosteroid (1.5 mL per level).

PRP: PRP preparation will occur at St. Joseph's Hospital using a standard 2-step centrifugation method. The Co-Investigator will draw 5-10cc of venous blood under sterile conditions (all patients) and subsequently centrifuge these samples at 200g for 10 minutes at room temperature. The plasma will then be separated from the sedimented erythrocytes and centrifuged again at 400g for 10 min to remove additional platelet-poor plasma. Finally, 1-2cc of PRP will be prepared for intra-articular injection. To maintain blinding, those in Group B will also have blood collection done, although their samples will not be injected.

Corticosteroid: 0.5 cc saline and 0.5cc of 10 mg/mL dexamethasone per facet joint (up to 6 mL total volume for 4 facet injections) will be prepared by the Principal Investigator or Co-Investigator.

Depending on randomization, the appropriate syringe will be delivered to the SJHC Pain Clinci interventional suite immediately after preparation. All injections will be performed by the same physician under fluoroscopic guidance at the same level(s) as the prior successful medial branch blocks. A small amount of contrast will be injected to ensure IA placement. It is recognized that IA placement may not be possible in every situation. It will be noted by the physician whether the injection is felt to be peri- or intra-articular.

Follow-up: Primary and secondary outcomes will be collected via phone or in person, pre-injection, and at 1, 3, and 6 months post-injection. If there is ongoing benefit ≥2 points on the NRS at 6 months, additional follow-up of primary and secondary outcomes at 9 and 12 months will be done.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Facetogenic neck pain at least 4/10 on NRS after whiplash injury
* At least 50% relief of familiar neck pain after dual cervical medial branch blocks

Exclusion Criteria:

* Suspected serious spinal pathology
* Fracture/dislocation at time of injury
* Nerve root compromise
* Spinal surgery or RFN in the past 12 months
* Prior corticosteroid cervical facet injection in past 6 months
* History of any uncontrolled mental health conditions
* Other contraindications to spinal injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-03-26 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline, 1, 3 and 6 months (+ 9 and 12 months) if at least an ongoing 2 point reduction at 6 months
  Numeric Rating Scale (NRS) rating from 0-10, 0 indicating no pain, and 10 indicating worst pain
Proportion attaining at least a 2 point reduction in pain on Numeric Rating Scale | 12 months
  Measured by Numeric Rating Scale questionnaire scores at Baseline, 1, 3 and 6 months (+ 9 and 12 months) if at least an ongoing 2 point reduction at 6 months. rating from 0-10, 0 indicating no pain, and 10 indicating worst pain
Proportion attaining 90% and 50% pain relief on Numeric Rating Scale | 12 months
  Measured by Numeric Rating Scale scores at Baseline, 1, 3 and 6 months (+ 9 and 12 months) if at least an ongoing 2 point reduction at 6 months. rating from 0-10, 0 indicating no pain, and 10 indicating worst pain
Time to return of at least 50% baseline pain on Numeric Rating Scale | 12 months
  Measured by Numeric Rating Scale questionnaire scores at baseline, 1, 3 and 6 months (+ 9 and 12 months) if at least an ongoing 2 point reduction at 6 months. rating from 0-10, 0 indicating no pain, and 10 indicating worst pain.

SECONDARY OUTCOMES:
Adverse Events | 12 months
  Including : increased pain, bleeding, infection, allergy, neurologic deficit, new hyperglycemia. Adverse events will be recorded through case report forms and reported to the principal investigator. Side effects will be assessed using standardized case report forms at each visit. Participants are encouraged to contact the coordinator to report any concerns.
Patient reported function in the presence of neck pain | 12 months
  Measured by the Neck Disability Index questionnaire, which is not a scale.
Patient's subjective satisfaction with the procedure | 12 months
  Measured by Modified MacNab criteria questionnaire at baseline, 1, 3 and 6 months (+ 9 and 12 months) if at least an ongoing 2 point reduction at 6 months. The MacNab criteria answers range from 1-4, 1 being excellent and 4 being poor.
Work Productivity and Activity | 12 months
  Change from baseline to end of study in the Work Productivity and Activity Questionnaire: Specific Health Impairment Version 2 (not a scale)
Self efficacy | 12 weeks.
  measured by self efficacy while performing daily activities in chronic WAD questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Eldon Loh, MD, Principal Investigator — St. Joseph's Healthcare London
Locations (1):
- St. Joseph's Health Care London, London, Ontario, Canada

REFERENCES:
- [Background] Carroll LJ, Holm LW, Hogg-Johnson S, Cote P, Cassidy JD, Haldeman S, Nordin M, Hurwitz EL, Carragee EJ, van der Velde G, Peloso PM, Guzman J; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Course and prognostic factors for neck pain in whiplash-associated disorders (WAD): results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S83-92. doi: 10.1097/BRS.0b013e3181643eb8. PMID 18204405
- [Background] Lim JW, Cho YW, Lee DG, Chang MC. Comparison of Intraarticular Pulsed Radiofrequency and Intraarticular Corticosteroid Injection for Management of Cervical Facet Joint Pain. Pain Physician. 2017 Sep;20(6):E961-E967. PMID 28934800
- [Background] Manchikanti L. Role of neuraxial steroids in interventional pain management. Pain Physician. 2002 Apr;5(2):182-99. PMID 16902669
- [Background] McDonald GJ, Lord SM, Bogduk N. Long-term follow-up of patients treated with cervical radiofrequency neurotomy for chronic neck pain. Neurosurgery. 1999 Jul;45(1):61-7; discussion 67-8. doi: 10.1097/00006123-199907000-00015. PMID 10414567
- [Background] Monfett M, Harrison J, Boachie-Adjei K, Lutz G. Intradiscal platelet-rich plasma (PRP) injections for discogenic low back pain: an update. Int Orthop. 2016 Jun;40(6):1321-8. doi: 10.1007/s00264-016-3178-3. Epub 2016 Apr 12. PMID 27073034
- [Background] Podd D. Platelet-rich plasma therapy: origins and applications investigated. JAAPA. 2012 Jun;25(6):44-9. doi: 10.1097/01720610-201206000-00009. No abstract available. PMID 22693884
- [Background] Quinn KP, Winkelstein BA. Detection of altered collagen fiber alignment in the cervical facet capsule after whiplash-like joint retraction. Ann Biomed Eng. 2011 Aug;39(8):2163-73. doi: 10.1007/s10439-011-0316-3. Epub 2011 May 3. PMID 21538155
- [Background] Teasell RW, McClure JA, Walton D, Pretty J, Salter K, Meyer M, Sequeira K, Death B. A research synthesis of therapeutic interventions for whiplash-associated disorder (WAD): part 5 - surgical and injection-based interventions for chronic WAD. Pain Res Manag. 2010 Sep-Oct;15(5):323-34. doi: 10.1155/2010/914358. PMID 21038011
- [Background] Wu J, Zhou J, Liu C, Zhang J, Xiong W, Lv Y, Liu R, Wang R, Du Z, Zhang G, Liu Q. A Prospective Study Comparing Platelet-Rich Plasma and Local Anesthetic (LA)/Corticosteroid in Intra-Articular Injection for the Treatment of Lumbar Facet Joint Syndrome. Pain Pract. 2017 Sep;17(7):914-924. doi: 10.1111/papr.12544. Epub 2017 Feb 22. PMID 27989008
- [Background] Barnsley L, Lord SM, Wallis BJ, Bogduk N. Lack of effect of intraarticular corticosteroids for chronic pain in the cervical zygapophyseal joints. N Engl J Med. 1994 Apr 14;330(15):1047-50. doi: 10.1056/NEJM199404143301504. PMID 8127332
- [Background] Falco FJ, Datta S, Manchikanti L, Sehgal N, Geffert S, Singh V, Smith HS, Boswell MV. An updated review of the diagnostic utility of cervical facet joint injections. Pain Physician. 2012 Nov-Dec;15(6):E807-38. PMID 23159977
- [Background] Hoy D, March L, Woolf A, Blyth F, Brooks P, Smith E, Vos T, Barendregt J, Blore J, Murray C, Burstein R, Buchbinder R. The global burden of neck pain: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1309-15. doi: 10.1136/annrheumdis-2013-204431. Epub 2014 Jan 30. PMID 24482302
- [Background] Le ADK, Enweze L, DeBaun MR, Dragoo JL. Current Clinical Recommendations for Use of Platelet-Rich Plasma. Curr Rev Musculoskelet Med. 2018 Dec;11(4):624-634. doi: 10.1007/s12178-018-9527-7. PMID 30353479
- [Background] Lord SM, Barnsley L, Wallis BJ, McDonald GJ, Bogduk N. Percutaneous radio-frequency neurotomy for chronic cervical zygapophyseal-joint pain. N Engl J Med. 1996 Dec 5;335(23):1721-6. doi: 10.1056/NEJM199612053352302. PMID 8929263
- [Background] MacVicar J, Borowczyk JM, MacVicar AM, Loughnan BM, Bogduk N. Cervical medial branch radiofrequency neurotomy in New Zealand. Pain Med. 2012 May;13(5):647-54. doi: 10.1111/j.1526-4637.2012.01351.x. Epub 2012 Mar 28. PMID 22458772
- [Background] Manchikanti L, Hirsch JA, Kaye AD, Boswell MV. Cervical zygapophysial (facet) joint pain: effectiveness of interventional management strategies. Postgrad Med. 2016 Jan;128(1):54-68. doi: 10.1080/00325481.2016.1105092. Epub 2015 Dec 10. PMID 26653406
- [Background] Persson M, Sorensen J, Gerdle B. Chronic Whiplash Associated Disorders (WAD): Responses to Nerve Blocks of Cervical Zygapophyseal Joints. Pain Med. 2016 Dec;17(12):2162-2175. doi: 10.1093/pm/pnw036. Epub 2016 Mar 27. PMID 28025352